CLINICAL TRIAL: NCT04520750
Title: VALO-2: A Multicenter, Phase 3b, Open-Label Treatment Extension Study Evaluating the Safety and Efficacy of PTX022 in the Treatment of Adults With Pachyonychia Congenita
Brief Title: VALO-2: Study Evaluating the Safety and Efficacy of PTX022 in the Treatment of Adults With Pachyonychia Congenita
Acronym: VALO-2
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Palvella Therapeutics, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: PALV-03
Record Dates: First submitted 2020-03-06; First posted 2020-08-20 (Actual); Last update posted 2024-08-29 (Actual); Status verified 2024-08

CONDITIONS: Pachyonychia Congenita
MeSH Terms: conditions — Pachyonychia Congenita

STUDY DESIGN:
Intervention Model Description: Open label
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- Open label treatment arm (Experimental): PTX-022 QTORIN
  Interventions: Drug: PTX-022

INTERVENTIONS:
Drug: PTX-022 — Safety and Efficacy of PTX-022 in the Treatment of Adults with Pachyonychia Congenita

SUMMARY:
VALO-2 is a multicenter, open-label extension (OLE) study enrolling patients with genotyped keratin mutations KRT6A, KRT6B and KRT16 who were previously treated with investigational PTX-022 during the VALO study. The purpose of the OLE study is to investigate long term exposure to investigational PTX-022 and evaluate safety and efficacy data. A sub-study is included to evaluate safety and efficacy of patients with genotyped keratin mutations of KRT6C and KRT17 not previously treated with investigational PTX-022.

ELIGIBILITY:
Key Inclusion Criteria:

* Adult patients 18 years or older,
* Previously completed the VALO protocol, or VALO-2 K6C/17 sub-study, and received meaningful benefit from investigational PTX-022 as determined by the clinician.

Key Exclusion Criteria:

* Any history of allergy or hypersensitivity to sirolimus, or sirolimus-like medications or to PTX-022

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 36 (Actual)
Dates: Start 2020-09-01 (Actual); Primary Completion 2021-06-30 (Actual); Study Completion 2022-12-15 (Actual)

PRIMARY OUTCOMES:
Incidence of Treatment-Emergent Adverse Events | 18 Months
Changes in vital sign measurements from baseline | 18 months
Changes in weight measurements from baseline | 18 months
Changes in clinical laboratory measurements from baseline | 18 months

SECONDARY OUTCOMES:
Patient Global Assessment of Activities Scale | 18 Months
Pain at its worst as assessed by NRS | 18 months
PROMIS Pain Interference Short 6A as assessed by likert scale | 18 months
PROMIS Physical Function as assessed by likert scale | 18 months
Patient Global Impression of Severity as assessed by likert scale | 18 months
Clinician Global Impression of Severity as assessed by likert scale | 18 months

CONTACTS AND LOCATIONS:
Locations (4):
- United States (4):
  - Arizona Research Center, Phoenix, Arizona
  - Stanford University, Palo Alto, California
  - Minnesota Clinical Study Center, Fridley, Minnesota
  - University of Utah, Murray, Utah